CLINICAL TRIAL: NCT05520853
Title: An Open, Single-arm, Multicenter Phase II Trial to Evaluate SBRT Combined With PD-1 Inhibitors and Thoracic Hyperthermia for Advanced Non-Small-Cell Lung Cancer
Brief Title: SBRT Combined With PD-1 Inhibitor and Thoracic Hyperthermia for Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bing Xia, Dr., First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-PT
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Stereotactic Body Radiation Therapy; PD-1 Inhibitor; Hyperthermia; NSCLC
MeSH Terms: conditions — Hyperthermia; Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT combined with PD-1 inhibitors and thoracic hyperthermia (Experimental): At least one lesion (primary or metastatic) was selected for SBRT treatment, and the radiotherapy dose of each lesion was 32Gy/4Fx. SBRT was combined with thoracic hyperthermia from the first fraction, and hyperthermia was performed 6 times, twice a week. PD-1 inhibitor was used on the second day after the completion of SBRT. The PD-1 inhibitor was administered at a dose of 200mg every time, every 3 weeks for 2 years (35 times total), or until the investigators deem that the patient need to discontinue the drug because of treatment-related toxicity or disease progression.
  Interventions: Radiation: SBRT combined with PD-1 inhibitors and thoracic hyperthermia

INTERVENTIONS:
Radiation: SBRT combined with PD-1 inhibitors and thoracic hyperthermia — At least one lesion (primary or metastatic) was selected for SBRT treatment, and the radiotherapy dose of each lesion was 32Gy/4Fx. SBRT was combined with thoracic hyperthermia from the first fraction, and hyperthermia was performed 6 times, twice a week. PD-1 inhibitor was used on the second day after the completion of SBRT. The PD-1 inhibitor was administered at a dose of 200mg every time, every 3 weeks for 2 years (35 times total), or until the investigators deem that the patient need to discontinue the drug because of treatment-related toxicity or disease progression.

SUMMARY:
The aim of this trial is to investigate the primary efficacy of SBRT combined with PD-1 inhibitor and thoracic hyperthermia in patients with EGFR, ALK, and ROS1 negative stage IV NSCLC patients who progressed after first-line treatment. At least one lesion (primary or metastatic) was selected for SBRT treatment, and the radiotherapy dose of each lesion was 32Gy/4Fx. SBRT was combined with thoracic hyperthermia from the first fraction, and hyperthermia was performed 6 times, twice a week. PD-1 inhibitor was used on the second day after the completion of SBRT. The PD-1 inhibitor was administered at a dose of 200mg every time, every 3 weeks for 2 years (35 times total), or until the investigators deem that the patient need to discontinue the drug because of treatment-related toxicity or disease progression. During the period, the overall response rate and toxicities were regularly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age≥18.
* 2.ECOG PS 0-1.
* 3.Histopathologically confirmed stage IV non-small-cell lung cancer.
* 4.EGFR/ALK/ROS-1 negetive.
* 5.Disease progression after first-line therapy including platinum chemotherapy, but not include PD-1/L1 inhibitors.
* 6.Subjects with brain metastases were eligible, but only if they had no neurologic symptoms or disease stable without systemic glucocorticoid.
* 7.At least one lesion with a diameter of 1-5cm which could be treated with SBRT at a dose of 32Gy/4Fx, and at least one lesion which could be measured other than SBRT (RECIST1.1); Lymph nodes can be used as independent measurable lesions or receive SBRT. Brain lesions should not be used as separate SBRT lesions or as measurable lesions.
* 8.The subjects did not had radiotherapy before.
* 9.The subjects did not currently need palliative radiotherapy at any part according to the researchers.
* 10.It was necessary for the subjects who underwent surgery to fully recover from the toxicity and complications caused by surgical intervention prior to treatment.
* 11.Subjects should provide appropriate biopsy specimens before and during treatment according to the clinical trial protocol.
* 12.Male or female subjects agree to contraception during the trial (surgical ligation or oral contraceptive/IUD + condom).
* 13.Life expectancy ≥ 3 months.
* 14.The organ function level meet the following standards one week before enrollment:

  ①Bone marrow: hemoglobin ≥80g/L, white blood cell count ≥4.0*10^9/L or neutrophil count ≥1.5*10^9/L, platelet count ≥100*10^9/L.

  ②Liver: Serum total bilirubin level ≤1.5 upper limit of normal (ULN), when serum total bilirubin level > 1.5 ULN, direct bilirubin level must be ≤ ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN.

  ③ Kidney: serum creatinine level < 1.5 ULN or creatinine clearance rate ≥ 50ml/min, urea nitrogen ≤ 200mg/L; Serum albumin ≥ 30g/L.
* 15. Subjects must be able to understand and voluntarily sign informed consent.

Exclusion Criteria:

* 1.Prior treatment with anti-PD-1 /L1 drugs or other investigational immunotherapy agent.
* 2.Subjects had prior radiotherapy.
* 3.Subjects had severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granuloma), etc.
* 4.Symptomatic interstitial lung disease or active infectious/noninfectious pneumonia.
* 5.Subjects had risk factors for bowel perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer, or other risk factors for bowel perforation.
* 6.History of other malignant tumors.
* 7.Subjects who have current infection, heart failure, heart attack, unstable angina, or unstable arrhythmia in the last 6 months.
* 8.Subjects with physical examination or clinical trial findings, or other uncontrolled conditions that the investigator believes may interfere with the outcome or increase the risk of treatment complications.
* 9.Subjects without platinum-based combination chemotherapy included as first-line treatment.
* 10.The pathology reports showed a mixture of small cell lung cancer components.
* 11.Lactating or pregnant women.
* 12.Congenital or acquired immunodeficiency diseases including human immunodeficiency virus (HIV), or a history of organ transplantation, allogeneic stem cell transplantation.
* 13.Known hepatitis B virus (HBV), hepatitis C virus (HCV), active pulmonary tuberculosis infections.
* 14.Subjects had cancer vaccines other vaccines within 4 weeks before treatment initiation. (Seasonal influenza vaccines are usually inactivated and are permitted, whereas intranasal preparations are usually live attenuated vaccines and therefore are not permitted)
* 15.Subjects who currently use other immune agents, chemotherapy agents, other investigational drugs or long-term cortisol therapy.
* 16.Subjects with mental illness, substance abuse, and social problems that affected compliance were not included in the study according to doctor's evaluation.
* 17.Allergic or contraindicated to PD-1 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 years
  The proportion of patients evaluated as complete response or partial response

SECONDARY OUTCOMES:
Incidence of treatment-related toxic effects | 2 years
  The proportion of treatment-related toxicity cases to the total number of evaluable cases assessed according to CTCAE 5.0 criteria
Objective response rate of non-irradiated lesions | 2 years
  The proportion of patients with non-irradiated lesions evaluated as complete response or partial response in the total enrolled patients
Overall response | 2 years
  The time span from the first day of enrollment until death from any cause
Progression free survival | 2 years
  The time span from the first day of enrollment until progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xia, MD, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Affiliated Hangzhou Cancer Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No